CLINICAL TRIAL: NCT04162808
Title: Development and Validation of a Full Course Bleeding Risk Assessment System for Antithrombotic Therapy of Acute Coronary Syndrome
Brief Title: Bleeding Risk Assessment System for Antithrombotic Therapy of ACS
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Beijing Anzhen Hospital (Other)
Collaborators: Peking Union Medical College Hospital (Other); Beijing Hospital (Other Government); Beijing Luhe Hospital (Other); Beijing Chao Yang Hospital (Other)
Responsible Party: Principal Investigator, Shao-Ping Nie, Professor of Medicine, Director, Emergency & Critical Care Center, Beijing Anzhen Hospital
Other Study IDs: 2018055X
Record Dates: First submitted 2019-11-12; First posted 2019-11-14 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Acute Coronary Syndrome
Keywords: bleeding; antithrombosis
MeSH Terms: conditions — Acute Coronary Syndrome; Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Antithrombotic therapy is the cornerstone of the management of patients with acute coronary syndrome (ACS), which result in lower risk of mortality and ischemic events. But, accompanied side effect of bleeding always causing worsens outcomes. Tools to evaluate risk/benefit ratio is useful in daily practice. The in-used scores, such as CRUSADE, are derived from retrospective studies, without all types of ACS and without long-term prediction. This project aims to establish a database of anti-thrombosis treatment and bleeding in five large centers in Beijing through the observational registry of ACS. With the database, establish a bleeding risk assessment system that can be used for all ACS patients and can predict the full course of antithrombotic treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age18-85 years old
2. Diagnosed ACS
3. Signed informed consent form

Exclusion Criteria:

1. Any active bleeding
2. Not tolerate to anti-thrombotic drugs
3. A planned elective surgical procedure that would necessitate an interruption in treatment with antiplatelet therapy in the next 6 months after enrollment
4. Patients who died of non-bleeding causes within 24 hours after admission
5. Noncardiac coexisting conditions that could limit life expectancy to less than 1 year
6. Pregnancy or lactation

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ACS patients
Sampling Method: Probability Sample
Enrollment: 6379 (Estimated)
Dates: Start 2018-01-04 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
The number of event of bleeding | 30 days
  The number of event of bleeding (BARC 2 to 5) within 30 days after enrollment
The number of event of bleeding | 1 year
  The number of event of bleeding (BARC 2 to 5) within 1 year after enrollment

SECONDARY OUTCOMES:
The number of event of bleeding | 30 days and 1 year
  The number of event of bleeding (BARC 1 to 5) within 30 days and 1year after enrollment
number of event of major adverse cardiovascular or cerebrovascular events | 30 days and 1 year
  number of event of major adverse cardiovascular or cerebrovascular events within 30 days and 1year after enrollment

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Anzhen Hospital, Beijing, China